CLINICAL TRIAL: NCT03244462
Title: Open Label, Randomized, Cross-over Study to Explore the Pharmacokinetics of BAY1834845 After Oral and Intravenous Dosing, Including Food Effect and Absolute Bioavailability (Part A), and to Investigate the Effect of BAY1834845 on the Pharmacokinetics of Orally Administered Methotrexate (Part B) in Healthy Male Subjects
Brief Title: Food Effect, Oral & Intravenous Pharmacokinetics and Absolute Bioavailability of BAY1834845 Including Drug-drug Interaction With Methotrexate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18387; 2016-004393-18 (EudraCT Number)
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — zabedosertib; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral BAY1834845 (Experimental): Study Part A, cross over sequence:
  1. single oral dose of BAY1834845
  2. single oral dose of BAY1834845 + i.v. BAY1834845
  3. single oral dose of BAY1834845 under fed conditions
  Interventions: Drug: BAY1834845
- Oral BAY1834845 + i.v. BAY1834845 (Experimental): Study Part A, cross over sequence:
  1. single oral dose of BAY1834845+ i.v. BAY1834845
  2. single oral dose of BAY1834845
  3. single oral dose of BAY1834845 under fed conditions
  Interventions: Drug: BAY1834845
- Oral Methotrexate (Experimental): Study part B, cross over sequence:
  1. single oral dose of methotrexate (MTX)
  2. single oral dose of MTX + single oral dose of BAY1834845
  Interventions: Drug: BAY1834845; Drug: Methotrexate
- Oral Methotrexate + oral BAY1834845 (Experimental): Study part B, cross over sequence:
  1. single oral dose of methotrexate (MTX) + single oral dose of BAY1834845
  2. single oral dose of MTX
  Interventions: Drug: BAY1834845; Drug: Methotrexate

INTERVENTIONS:
Drug: BAY1834845 — Single oral dose (IR [immediate release] tablets)
Drug: BAY1834845 — I.v. infusion of [13C6]-labeled BAY1834845
  Arms: Oral BAY1834845; Oral BAY1834845 + i.v. BAY1834845
Drug: Methotrexate — Single dose of commercially available MTX
  Arms: Oral Methotrexate; Oral Methotrexate + oral BAY1834845

SUMMARY:
This study is planned to explore the effect of food on the oral pharmacokinetics, the intravenous pharmacokinetics and the absolute bioavailability of BAY1834845. Furthermore, this study will investigate the effect of BAY1834845 on the pharmacokinetics of orally administered methotrexate in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male; healthy according to complete medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory tests as listed in the exclusion criteria given below.
* Age 18-50 years (inclusive) at the first screening visit.
* Body mass index: >=18 kg/m² and <=30 kg/m².
* Sexually active men must agree to practice adequate methods of contraception (protection).

This applies for the time period between signing of the informed consent form and up to 90 days after the last administration of the study drug(s).

Exclusion Criteria:

* Any contraindications for intake of BAY 1834845 or methotrexate, gastrointestinal, liver, renal, lung or cardiovascular disorders, malignant tumors, known severe allergies, known or suspected immunodeficiency
* Medication history: drugs known to induce/inhibit liver enzymes
* Smoking
* Clinically relevant findings in

  * physical
  * ECG, blood pressure
  * laboratory values
* Known hypersensitivity to study drug(s)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
AUC (Area under the concentration-versus-time curve from zero to infinity after single (first) dose) of BAY1834845 after oral administration of BAY1834845 to subjects in fed/fasted state | Multiple timepoints up to day 7
  in study part A
Maximum concentration attained (Cmax) of BAY1834845 after oral administration of BAY1834845 to subjects in fed/fasted state | Multiple timepoints up to day 7
  in study part A
Total body clearance (CL) of [13C6] BAY1834845 after intravenous administration | Multiple timepoints up to day 7
  in study part A
Volume of distribution at steady state (Vss) of [13C6] BAY1834845 after intravenous administration | Multiple timepoints up to day 7
  in study part A
Absolute oral bioavailability (F) of BAY1834845 in the fasted state | Multiple timepoints up to day 7
  in study part A
AUC of methotrexate in plasma in presence/absence of BAY1834845 | Multiple timepoints up to day 2
  in study part B
Cmax of methotrexate in plasma in presence/absence of BAY1834845 | Multiple timepoints up to day 2
  in study part B

SECONDARY OUTCOMES:
Frequency of Treatment Emergent Adverse Events (TEAEs) in part A | Up to 9 weeks
Severity of TEAEs in part A | Up to 9 weeks
Frequency of TEAEs in part B | Up to 6 weeks
Severity of TEAEs in part B | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- PRAHealthSciences, Groningen, Netherlands

REFERENCES:
- [Derived] Feldmuller M, Jodl SJ, Ploeger B, Wagenfeld A, Wiesinger H, Zollmann FS, Klein S, Zhang R, Rohde B, Hochel J. Zabedosertib, a novel interleukin-1 receptor-associated kinase-4 inhibitor, shows a favorable pharmacokinetic and safety profile across multiple phase 1 studies. Front Pharmacol. 2025 May 30;16:1521505. doi: 10.3389/fphar.2025.1521505. eCollection 2025. PMID 40520205